CLINICAL TRIAL: NCT05758870
Title: Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Brief Title: A Prospective Randomized Controlled Study Comparing the Clinical Effects of Surgical and Non-surgical Treatment of Low Rib Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Wu Weiming, Thoracic Surgery, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: 20220815
Record Dates: First submitted 2023-02-11; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Rib Fracture Multiple

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Research Group: surgical stabilization of low rib fracures by internal fixation
  Interventions: Procedure: surgical stabilization of low rib fratures
- Controls Group: conservative treatment of low rib fractures
  Interventions: Other: converstive treatment of low rib fratures

INTERVENTIONS:
Procedure: surgical stabilization of low rib fratures — surgical stabiliazation of rib fractures by internal fixation
  Groups: Research Group
Other: converstive treatment of low rib fratures — chest wall fixation band
  Groups: Controls Group

SUMMARY:
The purpose of this study is to explore the difference between the clinical effects of surgical and non-surgical treatment for patients with low rib fracture, and to explore whether SSRF has more clinical treatment advantages in patients with low rib fracture in a randomized, controlled and prospective manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest trauma only and unilateral low rib fractures Three rib fractures and more Displacement of the broken end of the fracture (bicortical fracture and not in the same line) Time from injury to hospital < 24 hours Age 18-70 ASA grade I-II Preoperative arterial oxygen partial pressure >60mmHg, carbon dioxide partial pressure <50mmHg The participate is volunteer in the study and sign the informed consent Pain score( Number Rating Scale, NRS) >5 under calm breathing

Exclusion Criteria:

* Difficult airway History of esophageal reflux Myasthenia gravis Coagulation disorders Gastrointestinal ulcer Gastrointestinal bleeding Anesthetic drugs allergy history Asthma Chronic obstructive pulmonary disease Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with multiple rib fractures combines with low rib fractures
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L | On the day of admission
  appraisal of life quality
EQ-5D-5L | 1 week after treatment
  appraisal of life quality
EQ-5D-5L | 2 weeks after treatment
  appraisal of life quality
EQ-5D-5L | 1 month after treatment
  appraisal of life quality
EQ-5D-5L | 3 months after treatment
  appraisal of life quality
EQ-5D-5L | 6 months after treatment
  appraisal of life quality

SECONDARY OUTCOMES:
Pain Score | On the day of admission
  Number Rating Score, NRS
Pain Score | 1 week after treatment
  Number Rating Score, NRS
Pain Score | 2 weeks after treanment
  Number Rating Score, NRS
Pain Score | 1 month after treatment
  Number Rating Score, NRS
Pain Score | 3 months after treatment
  Number Rating Score, NRS
Pain Score | 6 months after treatment
  Number Rating Score, NRS

OTHER OUTCOMES:
Atelectasis | On the day of admission
  CT scan show
Atelectasis | 1 week after treatment
  CT scan show
Atelectasis | 2 weeks after treanment
  CT scan show
Atelectasis | 1 month after treatment
  CT scan show
Atelectasis | 3 months after treatment
  CT scan show
Atelectasis | 6 months after treatment
  CT scan show
Pleural effusion | On the day of admission
  CT scan show
Pleural effusion | 1 week after treatment
  CT scan show
Pleural effusion | 2 weeks after treanment
  CT scan show
Pleural effusion | 1 months after treatment
  CT scan show
Pleural effusion | 3 months after treatment
  CT scan show
Pleural effusion | 6 months after treatment
  CT scan show
Mortality | On the day of admission
  death toll in each group
Mortality | 1 week after treatment
  death toll in each group
Mortality | 2 weeks after treanment
  death toll in each group
Mortality | 1 month after treatment
  death toll in each group
Mortality | 3 months after treatment
  death toll in each group
Mortality | 6 months after treatment
  death toll in each group
Length of hospital stay | the day from in the hospital to discharge
  time of hospitalization
Cost of treatment | the day from in the hospital to discharge
  total cost of hospitalization expense
Chest discomfort | On the day of admission
  chest tightness, foreign body sensation, numbness of surgical incision
Chest discomfort | 1 week after treatment
  chest tightness, foreign body sensation, numbness of surgical incision
Chest discomfort | 2 weeks after treanment
  chest tightness, foreign body sensation, numbness of surgical incision
Chest discomfort | 1 month after treatment
  chest tightness, foreign body sensation, numbness of surgical incision
Chest discomfort | 3 months after treatment
  chest tightness, foreign body sensation, numbness of surgical incision
Chest discomfort | 6 months after treatment
  chest tightness, foreign body sensation, numbness of surgical incision
Chronic pain | 3 months after treatment , 6 month after treatment
  pain for more than three months after surgery or trauma, NRS assessment
Chronic pain | 6 months after treatment
  pain for more than three months after surgery or trauma, NRS assessment
Duration of analgesic drug | the time of analgesic usement from first treat to the paitent do not use it anymore
  the time of analgesic usement from first treat to the paitent do not use it anymore
Total analgesic drug use | the time of analgesic usement from first treat to the paitent do not use it anymore
  total amont of analgesic usement from first treat to the paitent do not use it anymore
Lung function 1 | On the day of admission
  Forced vital capacity， FVC
Lung function 1 | 1 week after treatment
  Forced vital capacity， FVC
Lung function 1 | 2 weeks after treanment
  Forced vital capacity， FVC
Lung function 1 | 1 month after treatment
  Forced vital capacity， FVC
Lung function 1 | 3 months after treatment
  Forced vital capacity， FVC
Lung function 1 | 6 months after treatment
  Forced vital capacity， FVC
Lung function 2 | On the day of admission
  First second forced vital capacity，FEV1
Lung function 2 | 1 week after treatment
  First second forced vital capacity， FEV1
Lung function 2 | 2 weeks after treanment
  First second forced vital capacity， FEV1
Lung function 2 | 1 month after treatment
  First second forced vital capacity， FEV1
Lung function 2 | 3 months after treatment
  First second forced vital capacity， FEV1
Lung function 2 | 6 months after treatment
  First second forced vital capacity， FEV1